CLINICAL TRIAL: NCT00994578
Title: The COPE Trial: Communication in Oncologist-Patient Encounters
Brief Title: Intervention Study of Communication in Oncologist-Patient Encounters
Acronym: COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: Pro00013032; 2R01CA100387-06A1 (NIH)
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Advanced Cancer
Keywords: Advanced cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Internet Only (No Intervention): Patients assigned to the internet only group will enter the initial CHESS portal which will take them to a window displaying a standard web search engine and common cancer information sites. We will monitor their internet usage via logins to the CHESS portal.
- CHESS (Experimental): Participants in the CHESS arm will be given access to the University of Wisconsin CHESS website, modified specifically for this study. After being trained in usage of the site, they will use the available resources as desired without further input from the study team, except for technical support. The participant's usage of the site will be monitored.
  Interventions: Behavioral: CHESS
- COPE (Experimental): Participants in the COPE arm will receive training and access to the COPE patient intervention, an interactive web program based on Social Cognitive Theory that includes automated, tailored email reminders and encouragement prior to each visit, and access to the patient's audio-recorded conversations for review. The participant's usage of the site will be monitored.
  Interventions: Behavioral: COPE
- CHESS/COPE (Experimental): Participants in the CHESS+COPE arm will receive training in, and access to, both components on the CHESS website, with the accompanying levels of support. The participant's usage of the site will be monitored.
  Interventions: Behavioral: CHESS/COPE

INTERVENTIONS:
Behavioral: CHESS — Patients randomized to the CHESS intervention will be trained to access the website. After being trained in usage of the site, they will use the available resources as desired without further input from the study team, except for technical support
  Arms: CHESS
Behavioral: COPE — Participants in the COPE arm will receive training and access to the COPE patient intervention, an interactive web program based on Social Cognitive Theory that includes automated, tailored email reminders and encouragement prior to each of two oncologists visits over a maximum of a 9 month period, and access to the patient's audio-recorded conversations for review.
  Arms: COPE
Behavioral: CHESS/COPE — Participants in the CHESS/COPE arm will be given access to the University of Wisconsin CHESS modified specifically for this study. After being trained in usage of the site, they will use the available resources as desired and receive technical support. COPE arm will receive training and access to the COPE patient intervention an interactive web program based on Social Cognitive Theory that includes automated, tailored email reminders and encouragement prior to two oncologists visits over a maximum period of 9 months, and access to the patient's audio-recorded conversations for review.
  Arms: CHESS/COPE

SUMMARY:
The overall goal of this study is to improve communication between patients with advanced cancer and their oncologists. A web-based communication intervention will be delivered to patients to help them to express their negative emotions and elicit empathic responses from their oncologists.

The specific aims are to:

AIM 1: Develop a web-based intervention that trains patients with advanced cancer to express their emotional concerns to their oncologists and to request emotional support during clinical encounters.

AIM 2: Test whether this intervention can increase patient expression of emotional concerns and requests for emotional support, as well as improve patient affect by decreasing negative emotions.

DETAILED DESCRIPTION:
Patients will be recruited from the practices of participating oncologists; therefore, physicians will be enrolled prior to their patients. All medical, surgical and radiation oncology faculty and hematology/oncology fellows who see patients in the participating clinics will be eligible for the study. We will also enroll the mid-level providers (i.e., physician assistants and nurse practitioners) who work with many of these oncologists and any third party who comes to clinic with the enrolled patient.

Biweekly, we will present participating physicians with a list of potentially eligible patients (those with advanced disease) and ask them to identify those who should not be approached about study participation. Reasons to not approach include dementia or inappropriate disease staging. Identified patients will receive a letter from their treating oncologist inviting them to participate in the study about oncologist-patient communication. Patients who do not wish to be contacted about the study may call a toll-free number to opt out. If patients do not respond, a research assistant will contact them by telephone several days prior to their clinic visit, explain the study in detail, and obtain verbal consent to conduct a phone screener and baseline interview. It is necessary to conduct the screener and baseline survey prior to obtaining written consent so that staff may determine eligibility and then initiate study procedures at the upcoming clinic visit, if appropriate.

The baseline survey includes demographic information and several brief scales. Included in these is the Impact of Events Scale (IES) to determine level of distress, as the COPE study is interested in the subset of patients who are experiencing emotional difficulty with their cancer and may be amenable to support in this domain from their provider. The IES is scored from 0-44, with anything over 8 signifying at least mild levels of distress. Patients who score 10 or below will be excluded from the study. After completing the survey measures, arrangements will be made to meet patients in the clinic before their upcoming visit.

The research assistant will meet the patients in clinic, immediately prior to their next visit, and obtain written informed consent. After engaging in the informed consent process, the research assistant will place the audio recorder in the exam room, turn it on before the oncologist enters the room, exit the room, and then turn off the recorder at the end of the visit. S/he will not be present in the exam room during the visit. Subjects will complete a survey immediately after the visit to assess affect and quality of communication. Immediately after the visit, physicians will complete a very brief questionnaire to assess their perception of the subjects' distress and whether s/he talked about their distress.

Once research assistants determine that participating patients have an appointment with the same oncologist within 3 months, they will randomly assign subjects to one of four study arms (Control, CHESS, COPE, or CHESS+COPE), stratified by site and gender. Research assistants, equipped with laptop computers, will then introduce subjects to the intervention. For subjects in the Control arm, research assistants will use the intervention portal to review general Internet search tools (e.g., google). For subjects in the three intervention arms, research assistants will demonstrate the appropriately modified intervention website and ensure subjects' abilities to use it. Subjects will be provided written materials on the use of the website, and instructions will also be sent shortly afterward by email. The research assistant will call subjects within 7-14 days by phone and administer a 1-week follow-up survey to assess affect. This process will be repeated until staff record up to three clinic visits with the patient subject.

Staff will email and call patient subjects between clinic visits to remind them how to access the intervention website and answer technical questions. Also, research assistants will remind participants that a member of the study team will meet with them at their upcoming oncology appointments.

In the last post-visit call with patient subjects, staff will re-administer the IES. Once patients complete 3 audio-recorded visits, post-visits, and one-week follow-up interviews, study participation will be complete.

ELIGIBILITY:
Inclusion Criteria:

1. speak English;
2. have a diagnosis of advanced cancer (Stage IV or however defined for that disease group), metastatic disease, or refractory or recurrent illness;
3. have access to a telephone; and,
4. have regular access to a computer with broadband Internet service and an email account.

Exclusion Criteria:

1. incompetent for interview (documented diagnosis of active psychosis or dementia) or unable to provide informed consent as assessed by the interviewer;
2. hearing impaired or have a speech disorder;
3. physically impaired in such a way that precludes the use of a computer;
4. simply too sick to participate, and cannot realistically participate in the interview, as judged by the research assistant; or
5. does not have another appointment with an enrolled oncologist within three months.
6. has dial-up Internet service, or
7. does not meet IES Score.

While only patient subjects with advanced cancer will be eligible for randomization into one of the study arms, healthy volunteers (providers and third parties) will be enrolled in the study, too. Patients will be recruited from the practices of participating oncologists; therefore, physicians will be enrolled prior to their patients. All medical, surgical and radiation oncology faculty and hematology/oncology fellows who see patients in the participating clinics will be eligible for the study. We also will enroll the mid-level providers (i.e., physician assistants and nurse practitioners) who work with many of these oncologists and any third party (friends, family members) who comes to clinic with the enrolled patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2010-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Patient expression of emotion | Clinic Visits 2 and 3

SECONDARY OUTCOMES:
Patients randomized to the COPE only arm will have lower levels of negative affect and an increased number of requests for emotional support as compared to patients in the Internet only arm. | 9 months
Patients randomized to the CHESS only arm will have lower levels of negative affect as compared to patients in the Internet only arm. | 9 months
Patients randomized to the CHESS+COPE arm will have an increased number of expressions of emotional concerns and lower levels of negative affect as compared to patients in either the COPE only or CHESS only arms. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: James A Tulsky, MD, Principal Investigator — Duke University; Yael Schenker, MD, Principal Investigator — University of Pittsburgh; Kathryn Pollak, PhD, Study Director — Duke Health
Locations (2):
- United States (2):
  - Duke University Health System, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania